CLINICAL TRIAL: NCT04791150
Title: Rheumatologic Adverse Events and Immunotherapy in Oncology
Brief Title: Rheumatologic Adverse Events and Cancer Immunotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ONCOIMMUNO
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Oncology; Autoimmunity; Arthritis; Adverse Drug Event
MeSH Terms: conditions — Neoplasms; Autoimmune Diseases; Arthritis; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with cancer immunotherapy treatment (Experimental): All patients starting immunotherapy treatment will complete a questionnaire to identify rheumatological side effects, each time they come for treatment.
  Interventions: Other: Fill in a form

INTERVENTIONS:
Other: Fill in a form — Patient will have to fill in a form at each perfusion of immunotherapy to tell if they presents rheumatologic clinical signs

SUMMARY:
In this study, every patient with cancer who is going to be treated by immunotherapy will fill in a form. In this form, we try to determine if he presents rheumatologic complications of his immunotherapy. If the patient answers yes to one question on the form, the patient will be see in rheumatologic consultation to explore his clinical signs.

The number of patients referred in consultation thanks to this questionnaire will be compared to the number of patients who would have been spontaneously referred by the oncologist.

The aim of this questionnaire is to optimise the management of rheumatological effects secondary to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer needed to be treated by immunotherapy

Exclusion Criteria:

* Patient already treated by immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-07-07 (Estimated); Study Completion 2022-11-07 (Estimated)

PRIMARY OUTCOMES:
to determine whether a self-questionnaire completed by a patient treated with immunotherapy can identify more patients with rheumatological side effects related to this treatment, compared to the complaint reported by the patient to the oncologist | ONE YEAR
  number of patients referred to a rheumatology consultation thanks to the answers to the questionnaire compared to the number of patients referred to a consultation (from questionnaire and oncologist)

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No
NO IPD